CLINICAL TRIAL: NCT04406935
Title: Evaluation of the Safety and Efficacy of the NuEra Tight for Abdominal Circumference Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NuEra Tight-19-01
Record Dates: First submitted 2020-02-24; First posted 2020-05-29 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2020-02

CONDITIONS: Circumferential Reduction
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a Multi-arm, prospective, multi-center, baseline-controlled study, designed to evaluate the safety and efficacy of the NuEra Tight for circumferential reduction of the abdomen area at three different frequencies.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 475 KHz (Active Comparator): NuEra device treatment using 475 KHz
  Interventions: Device: treatment with the study device (NuEra)
- 1 MHz (Active Comparator): Arm 2: NuEra device treatment using 1 MHz
  Interventions: Device: treatment with the study device (NuEra)
- 2 MHz (Active Comparator): NuEra device treatment using 2 MHz
  Interventions: Device: treatment with the study device (NuEra)

INTERVENTIONS:
Device: treatment with the study device (NuEra) — Multi-arm, prospective, multi-center, baseline-controlled study:
  Arm 1: NuEra treatment using 475 KHz Arm 2: NuEra treatment using 1 MHz Arm 3: NuEra treatment using 2 MHz

SUMMARY:
Clinical study to evaluate the safety and efficacy of the NuEra Tight for circumferential reduction in the abdominal region within three treatment group

DETAILED DESCRIPTION:
The study design to evaluate the safety and efficacy of the NuEra Tight for circumferential reduction in the abdominal region within three treatment group. each group has a different radio-frequency. The study hypothesis is that NuEra Tight is safe and will cause a reduction in abdominal circumferential after treatment and at 12 week post last treatment within each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or Female, 18 to 65 years of age 2. Has visible fat bulges on the abdomen 3. Has a Body Mass Index (BMI) ≤ 30 4. Non-smoking for at least 6 months and willing to refrain from smoking for the duration of the study.

  5. Subject must agree to not undergo any other procedure(s) in the abdominal region during the study period.

  6. Subject who is willing to refrain from a change in diet/ exercise/medication regimen for the entire course of the study and to maintain his/her weight during the study within 5% of baseline weight measurement.

  7. Subject must agree to adhere to the follow-up schedule and study instructions.

  8. Subject must be able to read, understand and sign the Informed Consent Form. 9. Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.

  10. If the subject is a female and not pregnant or lactating, she must be either post-menopausal, surgically sterilized or using a medically acceptable form of birth control at least 3 months prior to enrolment (i.e oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence) and during the entire course of the study, and no plans to become pregnant.

Exclusion Criteria:

1. Subject had any type of prior cosmetic treatment to the target area within 12 months of study participation e.g., radiofrequency, cryolipolysis or light-based treatments.
2. Subject had any prior invasive cosmetic surgery to the target area, such as liposuction
3. Subject has scar tissue in and around the treatment area (i.e. cesarean-section or traumatic injury scar)
4. Subject has tattoo(s) that extend over a substantial portion of the treatment area
5. Subject is currently taking medications or supplements for weight-loss or metabolism support/enhancement or has a history of taking such medications or supplements within 3 months.
6. Has a pacemaker, internal defibrillator, implantable cardioverter-defibrillator, nerve stimulator implant, cochlear implant or any other electronically, magnetically or mechanically activated implant.
7. Has metal implant(s) within the body, such as surgical clips, plates and screws, intrauterine device (IUD), artificial heart valves or artificial joints.
8. History of diseases stimulated by heat, such as recurrent herpes zoster in the treatment area, unless treatment is conducted following a prophylactic regimen.
9. History of any disease or condition that could impair wound healing.
10. Infection, dermatitis, rash or other skin abnormality in the target area.
11. History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing
12. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, and abdominal aortic aneurysm
13. Significant concurrent illness, such as diabetes mellitus, hyperlipidemia, liver disease, HIV positive, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease, cardiovascular disease, peripheral vascular disease or pertinent neurological disorders.
14. History of skin disease in the treatment area or known epidermal or dermal disorders (particularly if involving collagen or microvascularity)
15. Severe skin laxity in the treatment area
16. Extensive collection of visceral adipose tissue or abdominal wall diastasis or hernia on physical examination
17. Obesity ≥30 BMI
18. Diagnosed or documented immune system disorders.
19. Currently undergoing systemic chemotherapy or radiation treatment for cancer, or history of treatment in the target area within 3 months of study participation.
20. Participation in a clinical trial of another device or drug within 6 months of study participation, or during the study period.
21. Pregnant or currently breastfeeding.
22. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.
23. Known allergy to general and/or topical anesthetic

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Reduction in abdominal circumference | one month
  Change in abdominal circumference in cm

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Skincare Physicians, Chestnut Hill, Massachusetts
  - Dermatology and Laser Surgery Center of New York, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided